CLINICAL TRIAL: NCT03243734
Title: A Prospective Single Arm Multicenter Study Evaluating the Effects of Spray Cryotherapy in Patients With Persistent Local Esophageal Cancer
Brief Title: trūFreeze® Palliative Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Endoscopy Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 017
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
Keywords: spray cryotherapy; quality of life; symptom reduction; esophageal malignancies; liquid nitrogen; ablation
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- trūFreeze® System spray cryotherapy (Experimental): trūFreeze® System spray cryotherapy as clinically indicated for symptom relief
  Interventions: Device: trūFreeze® System spray cryotherapy

INTERVENTIONS:
Device: trūFreeze® System spray cryotherapy — Subjects where trūFreeze® System spray cryotherapy is performed

SUMMARY:
Prospective, open label, non-controlled single arm, multi-center study The primary objective is to study the effects of the trūFreeze® Spray Cryotherapy System in a population of subjects who have been diagnosed with persistent local esophageal cancer and who are not surgical candidates or have completed or declined systemic therapy.

DETAILED DESCRIPTION:
The use of cryotherapy delivered with the trūFreeze® System via noncontact spray ablates the cancer cells while allowing adjacent normal tissue to regenerate. When the liquid nitrogen is delivered to the malignant lesion the cancer cells undergo ablation induced by intracellular water being frozen in place such that ice crystals are formed. These ice crystals aggregate quickly causing immediate intracellular energy producing organelles to be destroyed leading to a non-viable cell. Subsequent tumor sloughing and absorption of apoptotic cells occurs with a subsequent debulking of the tumor mass. Normal tissue will regenerate as re-epithelialization occurs. The extreme cold of -196 degrees Celsius or a "hard freeze" leads to more extensive primary cell death over a shorter freeze time as compared to cryoprobes. A reduction of overall tumor obstruction in the esophageal lumen can reduce symptoms of dysphagia, delay the time until stent is needed, provide palliative care for patients for whom additional tri-modal therapies are not an option, and may increase quality of life in esophageal cancer patients. The studies conducted to date have provided documentation of the safety and effectiveness of spray cryotherapy (SCT) when used for malignancies in the esophagus. Measures of dysphagia relief have been described in peer reviewed literature. This study aims to provide much needed HRQOL information as well as additional tumor characteristics before and after SCT. A cohort of patients with locally persistent esophageal cancer will be studied in up to twelve (12) centers in the United States to provide important HRQOL data and more a comprehensive understanding of clinical tumor response post SCT. In the proposed study, the trūFreeze® System spray cryotherapy procedure will be performed during endoscopy. Each SCT procedure will be performed endoscopically at clinically indicated intervals of 6 weeks +/- 3 weeks. Total procedure dosimetry will be delivered at the discretion of the Investigator based on tumor location and patient tolerability. After each procedure at defined intervals, patients will be contacted and QOL symptom related information will be collected. If at any point an Investigator determines that a subject is not a candidate for further spray cryotherapy or is unable to tolerate additional procedures, they will be contacted via telephone to ascertain HRQOL information. Subject participation will last up to two years or until death

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 18 to 89 years of age.
* Subject is able to read, understand, and sign a written Informed Consent to participate in the study.
* Subject has persistent esophageal cancer with local luminal involvement and who is not a surgical candidate or has completed or declined systemic therapy.
* Subject is able to tolerate endoscopy

Exclusion Criteria:

* Subject is pregnant, nursing, or planning to get pregnant during study duration.
* Subjects with an esophageal stent in situ at the time of study enrollment
* Subject, as deemed by treating investigator has contraindication to endoscopy or Spray Cryotherapy Procedure.
* Subject has received radiation within the past 6 weeks
* Subject has received chemotherapy within the past 2 weeks Subject has received immunotherapy within 30 days
* Subject has participated in another clinical study for systemic therapy within 6 weeks of baseline.
* Subject has had previous Spray Cryotherapy for esophageal cancer.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline EORTC at 14 days post cryotherapy procedure | 14 days post spray cryotherapy
  Validated Cancer Specific Quality of Life Questionnaire
Change from baseline dysphagia scale at 14 days post cryotherapy procedure | 14 days post spray cryotherapy
  Dysphagia Severity Scale

SECONDARY OUTCOMES:
Time to additional interventional procedure(s) other than spray cryotherapy (e.g. stent placement) | up to 2 years post SCT procedure
  baseline to procedure other than spray cryotherapy
Overall Survival | up to 2 years post SCT procedure
  SCT to death
Mean change in the amount of residual tumor from baseline to follow-up cryospray delivery session | up to 2 years post SCT procedure
  Describe changes in tumor

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Shaheen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (10):
- United States (10):
  - Cancer Treatment Centers of America Western Regional Medical Center, Goodyear, Arizona
  - University of California at Irvine, Orange, California
  - Emory University, Atlanta, Georgia
  - Parkview Comprehensive Cancer Center, Fort Wayne, Indiana
  - Spectrum Health, Grand Rapids, Michigan
  - Dartmouth-Hotchcock Medical Center, Lebanon, New Hampshire
  - North Shore-Long Island Jewish Medical Center, Manhasset, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No